CLINICAL TRIAL: NCT04784754
Title: A Pilot Placebo-controlled Randomized Double-blind Trial of Melatonin in Outpatients With COVID-19 Infection
Brief Title: Dose-Ranging Study to Assess the Safety and Efficacy of Melatonin in Outpatients Infected With COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of subject enrollment
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Margarita L. Dubocovich, PhD, SUNY Distinguished Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UBMELCOVID19-P; UL1TR001412 (NIH)
Record Dates: First submitted 2021-02-22; First posted 2021-03-05 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
Keywords: Melatonin; COVID-19; outpatient; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Melatonin; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Placebo-controlled randomized double-blind trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo capsules will be prepared using hypromellose capsules, filled using microcrystalline cellulose. This is the same excipient used in the preparation of the interventional drug. Placebo will be administered orally three times a day for 14 days in the same regimen used for the intervention.
  Interventions: Drug: Placebo
- Melatonin 3 mg (Experimental): Melatonin capsules will be prepared using hypromellose capsules containing 3 mg of the active component and identical excipient (Microcrystalline Cellulose) used in the placebo preparation. Melatonin will be administered orally three times a day for 14 days.
  Interventions: Drug: Melatonin
- Melatonin 30 mg (Experimental): Melatonin capsules will be prepared using hypromellose capsules containing 30 mg of the active component and identical excipient (Microcrystalline Cellulose) used in the placebo preparation. Melatonin will be administered orally three times a day for 14 days.
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — Melatonin capsules will be prepared using hypromellose capsules containing 3 mg or 30 mg of the active component and identical excipient (Microcrystalline Cellulose) used in the placebo preparation. Melatonin will be administered orally three times a day for 14 days.
  Other Names: 5-methoxy-N-acetyl tryptamine
  Arms: Melatonin 3 mg; Melatonin 30 mg
Drug: Placebo — Placebo capsules will be prepared using hypromellose capsules, filled using microcrystalline cellulose. This is the same excipient used in the preparation of the interventional drug. Placebo will be administered orally three times a day for 14 days in the same regimen used for the intervention.
  Other Names: Microcrystalline Cellulose
  Arms: Placebo

SUMMARY:
A pilot placebo-controlled randomized double-blind trial of Melatonin in outpatients with COVID-19 infection to evaluate Safety, Efficacy and Dose-ranging.

DETAILED DESCRIPTION:
Studies have shown in the blood of patients with COVID-19 there was a marked increase in the cytokines and chemokines interleukin 1β (IL-1β), interferon-γ (IFN-γ), interferon-inducible protein 10 (IP-10), monocyte chemoattractant protein 1 (MCP-1) and interleukin-4 (IL-4). Consequently, treatments that reduce cytokine/chemokine production that result in a less severe course of disease could be potentially beneficial. Melatonin, a pineal hormone, has been shown to have anti-inflammation, anti-oxidation and immune enhancing features. In multiple animal models of lung injury, Melatonin supplementation has been shown to decrease the number of inflammatory cells, reduce the levels of the cytokines IL-4, IL-5, IL-13 and TNF-a and reduce nitric oxide and hydroxyl radical concentrations. We propose a dose ranging pilot study to assess the safety and efficacy of melatonin in reducing hospitalization in COVID-19 patients with mild-moderate disease. A total of 50 participants will be randomized to the intervention arm (melatonin: 3 mg, or 30 mg three times a day for 14 days) or control arm (placebo) in a 2:2:1 fashion using a permuted block randomization scheme. Analyses will be performed with a focus on estimation of specific clinically important parameters, including safety and preliminary evidence of activity, for planning of a subsequent definitive comparative trial designed to fully assess efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female adult ≥18 years of age at time of enrollment.
2. Women of childbearing potential must agree to use at least one primary form of contraception for the duration of the study.
3. Positive testing for COVID-19 infection by standard RT-PCR assay or equivalent test.
4. Meets criteria for mild or moderate COVID-19 disease
5. Subject provides written informed consent prior to initiation of any study procedures.
6. Understands and agrees to comply with planned study procedures.
7. Agrees to the collection and storage of saliva samples per protocol.
8. Subject can provide an emergency contact who the study team can contact in case the subject is not reachable on any of the study visits.

Exclusion Criteria:

1. Severe (eGFR<30 ml/min) and moderate (eGFR 30-60 ml/min) chronic kidney disease or requiring dialysis
2. Severe hepatic insufficiency defined as one or more of the following: Cirrhosis diagnosis, Serum ALT > 3x ULN or Alkaline phosphatase >3x ULN or bilirubin >2x ULN in the absence of Gilbert's or hemolysis, Uncontrolled acute or chronic liver disease (e.g. acute hepatitis A, unstable autoimmune hepatitis)
3. Pregnancy or breast feeding.
4. History of a seizure disorder.
5. Patient is taking Fluvoxamine, Capmatinib, Ciprofloxacin (Systemic), Deferasirox, Givosiran, Methoxsalen (Systemic), Mexiletine, Rucaparib, Stiripentol, Thiabendazole, Vemurafenib, Methoxsalen, Sodium oxybate or Echinacea.
6. Allergy to the study medication
7. Currently taking melatonin
8. Currently taking high dose (>500 mg/day) Vitamin C.
9. Meets criteria for Severe or Critical COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative Incidence of Treatment-Emergent Adverse Events | 42 days
  Evaluate the incidence of serious adverse effects and discontinuation secondary to toxicity through 42 days of follow-up as compared to the control arm as assessed by: Cumulative incidence of serious adverse events (SAEs), Cumulative incidence of Grade 3 and 4 adverse events (AEs), Discontinuation or temporary suspension of the investigational medication (for any reason).

SECONDARY OUTCOMES:
Incidence of COVID-19 related hospitalization | 42 days
  Incidence of COVID-19 related hospitalization at 42 days
COVID-19 related symptoms | 42 days
  COVID-19 related symptoms as self-reported and on interview.
Rate of resolution of COVID-19 related symptoms | up to 42 days
  Change from baseline (day 1) as assessed to days 3, 7, 14, 28 and 42
Mortality | 42 days
  42-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Margarita L Dubocovich, PhD, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aliasgharzadeh A, Farhood B, Amini P, Saffar H, Motevaseli E, Rezapoor S, Nouruzi F, Shabeeb DH, Eleojo Musa A, Mohseni M, Moradi H, Najafi M. Melatonin Attenuates Upregulation of Duox1 and Duox2 and Protects against Lung Injury following Chest Irradiation in Rats. Cell J. 2019 Oct;21(3):236-242. doi: 10.22074/cellj.2019.6207. Epub 2019 Jun 15. PMID 31210428
- [Background] Andersen LP, Gogenur I, Rosenberg J, Reiter RJ. The Safety of Melatonin in Humans. Clin Drug Investig. 2016 Mar;36(3):169-75. doi: 10.1007/s40261-015-0368-5. PMID 26692007
- [Background] Bazyar H, Gholinezhad H, Moradi L, Salehi P, Abadi F, Ravanbakhsh M, Zare Javid A. The effects of melatonin supplementation in adjunct with non-surgical periodontal therapy on periodontal status, serum melatonin and inflammatory markers in type 2 diabetes mellitus patients with chronic periodontitis: a double-blind, placebo-controlled trial. Inflammopharmacology. 2019 Feb;27(1):67-76. doi: 10.1007/s10787-018-0539-0. Epub 2018 Oct 16. PMID 30328031
- [Background] Chen CF, Wang D, Reiter RJ, Yeh DY. Oral melatonin attenuates lung inflammation and airway hyperreactivity induced by inhalation of aerosolized pancreatic fluid in rats. J Pineal Res. 2011 Jan;50(1):46-53. doi: 10.1111/j.1600-079X.2010.00808.x. Epub 2010 Oct 22. PMID 20964706
- [Background] Cheung CY, Poon LL, Ng IH, Luk W, Sia SF, Wu MH, Chan KH, Yuen KY, Gordon S, Guan Y, Peiris JS. Cytokine responses in severe acute respiratory syndrome coronavirus-infected macrophages in vitro: possible relevance to pathogenesis. J Virol. 2005 Jun;79(12):7819-26. doi: 10.1128/JVI.79.12.7819-7826.2005. PMID 15919935
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Kim JY, Lee YD, Kim BJ, Kim SP, Kim DH, Jo KJ, Lee SK, Lee KH, Baik HW. Melatonin improves inflammatory cytokine profiles in lung inflammation associated with sleep deprivation. Mol Med Rep. 2012 May;5(5):1281-4. doi: 10.3892/mmr.2012.814. Epub 2012 Feb 29. PMID 22377793
- [Background] Law HK, Cheung CY, Ng HY, Sia SF, Chan YO, Luk W, Nicholls JM, Peiris JS, Lau YL. Chemokine up-regulation in SARS-coronavirus-infected, monocyte-derived human dendritic cells. Blood. 2005 Oct 1;106(7):2366-74. doi: 10.1182/blood-2004-10-4166. Epub 2005 Apr 28. PMID 15860669
- [Background] Pedreira PR, Garcia-Prieto E, Parra D, Astudillo A, Diaz E, Taboada F, Albaiceta GM. Effects of melatonin in an experimental model of ventilator-induced lung injury. Am J Physiol Lung Cell Mol Physiol. 2008 Nov;295(5):L820-7. doi: 10.1152/ajplung.90211.2008. Epub 2008 Sep 19. PMID 18805959
- [Background] Peng Z, Zhang W, Qiao J, He B. Melatonin attenuates airway inflammation via SIRT1 dependent inhibition of NLRP3 inflammasome and IL-1beta in rats with COPD. Int Immunopharmacol. 2018 Sep;62:23-28. doi: 10.1016/j.intimp.2018.06.033. Epub 2018 Jun 30. PMID 29990691
- [Background] Sanchez-Lopez AL, Ortiz GG, Pacheco-Moises FP, Mireles-Ramirez MA, Bitzer-Quintero OK, Delgado-Lara DLC, Ramirez-Jirano LJ, Velazquez-Brizuela IE. Efficacy of Melatonin on Serum Pro-inflammatory Cytokines and Oxidative Stress Markers in Relapsing Remitting Multiple Sclerosis. Arch Med Res. 2018 Aug;49(6):391-398. doi: 10.1016/j.arcmed.2018.12.004. Epub 2018 Dec 27. PMID 30595364
- [Background] Shang Y, Xu SP, Wu Y, Jiang YX, Wu ZY, Yuan SY, Yao SL. Melatonin reduces acute lung injury in endotoxemic rats. Chin Med J (Engl). 2009 Jun 20;122(12):1388-93. PMID 19567158
- [Background] Shin IS, Park JW, Shin NR, Jeon CM, Kwon OK, Kim JS, Kim JC, Oh SR, Ahn KS. Melatonin reduces airway inflammation in ovalbumin-induced asthma. Immunobiology. 2014 Dec;219(12):901-8. doi: 10.1016/j.imbio.2014.08.004. Epub 2014 Aug 10. PMID 25161126
- [Background] Wang S, Zhao Z, Feng X, Cheng Z, Xiong Z, Wang T, Lin J, Zhang M, Hu J, Fan Y, Reiter RJ, Wang H, Sun D. Melatonin activates Parkin translocation and rescues the impaired mitophagy activity of diabetic cardiomyopathy through Mst1 inhibition. J Cell Mol Med. 2018 Oct;22(10):5132-5144. doi: 10.1111/jcmm.13802. Epub 2018 Jul 31. PMID 30063115
- [Background] Wu GC, Peng CK, Liao WI, Pao HP, Huang KL, Chu SJ. Melatonin receptor agonist protects against acute lung injury induced by ventilator through up-regulation of IL-10 production. Respir Res. 2020 Mar 6;21(1):65. doi: 10.1186/s12931-020-1325-2. PMID 32143642
- [Background] Wu WS, Chou MT, Chao CM, Chang CK, Lin MT, Chang CP. Melatonin reduces acute lung inflammation, edema, and hemorrhage in heatstroke rats. Acta Pharmacol Sin. 2012 Jun;33(6):775-82. doi: 10.1038/aps.2012.29. Epub 2012 May 21. PMID 22609835
- [Background] Zhao X, Sun J, Su W, Shan H, Zhang B, Wang Y, Shabanova A, Shan H, Liang H. Melatonin Protects against Lung Fibrosis by Regulating the Hippo/YAP Pathway. Int J Mol Sci. 2018 Apr 9;19(4):1118. doi: 10.3390/ijms19041118. PMID 29642520
- [Background] Zhang R, Wang X, Ni L, Di X, Ma B, Niu S, Liu C, Reiter RJ. COVID-19: Melatonin as a potential adjuvant treatment. Life Sci. 2020 Jun 1;250:117583. doi: 10.1016/j.lfs.2020.117583. Epub 2020 Mar 23. PMID 32217117